CLINICAL TRIAL: NCT04183491
Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: Clinical Study 3 - Interferon Beta-1A and Peginterferon Beta-1A
Brief Title: Pharmacodynamic Biomarkers to Support Biosimilar Development: Interferon Beta-1A Products
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SCR-008
Record Dates: First submitted 2019-11-27; First posted 2019-12-03 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subjects; Pharmacokinetics; Pharmacodynamics
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Interferon beta-1a; peginterferon beta-1a

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of three dose groups (low, intermediate, and high) of each drug (interferon beta-1a and peginterferon beta-1a) or placebo
Who Masked: Participant, Investigator
Masking Description: The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
  Subjects and staff will be blinded to treatment assignment during confinement, but route of administration will not be blinded. The blind will be maintained through a randomization schedule held by the dispensing pharmacist. Subjects and staff will be informed of a subject's end of study day when discharged from confinement. Subjects and staff will not be informed of the specific treatment arm assignment. The clinical research nurse will administer the subcutaneous study drug in unit dose containers that are not transparent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm A: Interferon beta-1a low dose (Experimental): Single dose of interferon beta-1a 7.5 µg intramuscular (IM)
  Interventions: Biological: Interferon beta-1a
- Arm B: Interferon beta-1a intermediate dose (Experimental): Single dose of interferon beta-1a 15 µg IM
  Interventions: Biological: Interferon beta-1a
- Arm C: Interferon beta-1a high dose (Experimental): Single dose of interferon beta-1a 30 µg IM
  Interventions: Biological: Interferon beta-1a
- Arm D: Peginterferon beta-1a low dose (Experimental): Single dose of peginterferon beta-1a 31.25 µg subcutaneous (SC)
  Interventions: Biological: Peginterferon beta-1a
- Arm E: Peginterferon beta-1a intermediate dose (Experimental): Single dose of peginterferon beta-1a 62.5 µg SC
  Interventions: Biological: Peginterferon beta-1a
- Arm F: Peginterferon beta-1a high dose (Experimental): Single dose of peginterferon beta-1a 125 µg SC
  Interventions: Biological: Peginterferon beta-1a
- Arm G: Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Interferon beta-1a — Interferon beta-1a 7.5 µg administered IM
  Arms: Arm A: Interferon beta-1a low dose
Biological: Interferon beta-1a — Interferon beta-1a 15 µg administered IM
  Arms: Arm B: Interferon beta-1a intermediate dose
Biological: Interferon beta-1a — Interferon beta-1a 30 µg administered IM
  Arms: Arm C: Interferon beta-1a high dose
Biological: Peginterferon beta-1a — Peginterferon beta-1a 31.25 µg administered SC
  Arms: Arm D: Peginterferon beta-1a low dose
Biological: Peginterferon beta-1a — Peginterferon beta-1a 62.5 µg administered SC
  Arms: Arm E: Peginterferon beta-1a intermediate dose
Biological: Peginterferon beta-1a — Peginterferon beta-1a 125 µg administered SC
  Arms: Arm F: Peginterferon beta-1a high dose
Biological: Placebo — Placebo (administered either IM or SC)
  Arms: Arm G: Placebo

SUMMARY:
This study is designed to assess pharmacokinetics and pharmacodynamics of interferon beta-1a and peginterferon beta-1a across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 84 healthy subjects assigned to one of three dose groups (low, intermediate, and high) of each drug (interferon beta-1a and peginterferon beta-1a) or placebo.

DETAILED DESCRIPTION:
This study is designed to assess pharmacokinetics and pharmacodynamics of interferon beta-1a and peginterferon beta-1a across an appropriate dose range to inform clinical trial operating characteristics for future clinical pharmacology pharmacodynamics similarity studies.

This is a randomized, placebo-controlled, single-dose, parallel arm study in 84 healthy subjects assigned to one of three dose groups (low, intermediate, and high) of each drug (interferon beta-1a and peginterferon beta-1a) or placebo. Interferon beta-1a doses are 7.5, 15, and 30 µg. Peginterferon beta-1a doses are 31.25, 62.5, and 125 µg. Each arm will include 12 subjects (6 male and 6 female).

Subjects will be admitted for treatment on day -1 and receive a single dose of study drug or placebo on day 1. Depending on the treatment arm, subjects will remain in confinement for 7 days (interferon beta-1a) or 14 days (peginterferon beta-1a and placebo).

Blood samples (approximately 5 mL per sample) will be collected for determination of plasma concentrations for study drug and neopterin levels. Additional blood samples will be collected for determination of lipids (5 mL per sample; pharmacodynamic measure) and exploratory proteomics analyses (5 mL per sample).

Safety evaluations will include adverse event (AE) monitoring, vital sign measurements, and physical examinations. All AEs reported by the subject or observed by the investigator or clinical research unit (CRU) staff will be recorded. Any AE reported after the informed consent is signed and before study drug application will be recorded as medical history.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 55 years of age, inclusive, who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and drugs of abuse at screening and Check-in (Day -1).
5. Female subjects must be of non-childbearing potential or, if they are of childbearing potential, they must: 1) have been strictly abstinent for 1 month before Check in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 2) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from at least 1 month before Check in (Day -1) until at least 1 month after the last application of study drug.
6. Female subjects must not be pregnant or lactating before enrollment in the study.
7. Male subjects must agree to practice 1 highly effective method of birth control (as determined by the investigator or designee) from at least 1 month before Check-in (Day -1) until at least 1 month after the end of study
8. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Subject has had previous exposure to the biologic Avonex or Plegridy.
2. Subject is anemic (i.e., with Hct or Hgb considered clinically significant by Investigator or chronic history of anemia) or has any chronic condition(s) that may impact blood sample collection.
3. Subject has a history of asthma.
4. Subject has a history of anaphylaxis from environmental exposures such as peanuts or bee stings.
5. Subject has an allergic history that includes urticaria, angioedema or respiratory coughing or bronchospasm.
6. Subject has a history of severe local reactions or generalized erythema from skin allergen testing.
7. Subject has used any prescription or nonprescription drugs (including aspirin or NSAIDs and excluding oral contraceptives and acetaminophen) within 14 days or 5 half-lives (whichever is longer) or complementary and alternative medicines within 28 days before the first dose of study drug.
8. Subjects are currently participating in another clinical study of an investigational drug or are have been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of the compound.
9. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks of Screening.
10. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 hours of dosing. Subjects must refrain from ingesting these throughout the study.
11. Subject has any underlying disease or surgical or medical condition (e.g., cancer, human immunodeficiency virus [HIV], severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study. This includes subjects with any underlying medical conditions that put subjects at higher risk for coronavirus disease of 2019 (COVID-19) complications. Per current Center for Disease Control and Prevention (CDC) recommendations, this includes:

    * People with chronic lung disease or moderate to severe asthma
    * People who have serious heart conditions
    * People who are immunocompromised
    * Many conditions can cause a person to be immunocompromised, including cancer treatment, smoking, bone marrow or organ transplantation, immune deficiencies, poorly controlled HIV, and prolonged use of corticosteroids and other immune weakening medications
    * People with severe obesity (BMI of 40 or higher)
    * People with diabetes
    * People with chronic kidney disease undergoing dialysis
    * People with liver disease
12. Subject has any signs or symptoms that are consistent with COVID-19. Per current CDC recommendations, this includes subjects with the symptoms of cough or shortness of breath or difficulty breathing, or at least two of the following symptoms: fever, chills, repeated shaking with chills, muscle pain, headache, sore throat or new loss of taste/smell. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
13. Subject tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a molecular diagnostic test performed prior to admission.
14. Subject has been diagnosed with any autoimmune disease or other chronic inflammatory disease.
15. Subject has been diagnosed with depression, suicidal ideation or psychosis.
16. Subject has been diagnosed with congestive heart failure.
17. Subject has been diagnosed with seizures of any type.
18. Subject has known or suspected allergies or sensitivities to any study drug.
19. Subject has clinical laboratory test results (hematology, serum chemistry lipid panel and comprehensive metabolic panel) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
20. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
21. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as a part of manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as any eventual publications.
Supporting Information: Study Protocol, SAP
Time Frame: February, 2022. Materials will be available indefinitely.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose | Arm G: Placebo
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 11 | 12 | 12 | 11 | 12
Not Completed | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose | Arm G: Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (8.6) | 35.1 (9.7) | 38.3 (10.9) | 37.7 (12.7) | 31.9 (11.1) | 35.5 (8.0) | 36.9 (10.6) | 35.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 5 | 5 | 4 | 4 | 32
  Male | 7 | 7 | 8 | 7 | 7 | 8 | 8 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 3 | 1 | 1 | 1 | 10
  Not Hispanic or Latino | 9 | 11 | 12 | 9 | 11 | 11 | 11 | 74
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 8 | 7 | 6 | 8 | 4 | 6 | 41
  White | 8 | 3 | 4 | 6 | 4 | 8 | 5 | 38
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 84
Body weight [Mean (Standard Deviation); unit: kg] | 73.5 (11.4) | 72.7 (12.2) | 80.0 (14.5) | 78.5 (10.7) | 76.3 (13.2) | 76.3 (10.9) | 79.3 (9.1) | 76.7 (11.7)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.5 (2.3) | 25.9 (2.7) | 27.0 (3.0) | 26.2 (3.2) | 27.0 (2.6) | 25.6 (2.5) | 27.1 (2.4) | 26.2 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Area Under Effect Curve (AUEC) for Neopterin for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of standard pharmacodynamic (PD) metric (AUEC [baseline subtracted]) for neopterin at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: 0, 1, 3, 6, 8, 16, 24, 32, 40, 48, 72, hours post-dose; once daily from Day 4 onwards until 7 days post-dose for Interferon Beta-1a treatment arms (Arms A, B and C) and 14 days post-dose for Peginterferon Beta-1a treatment arms (Arms D, E, and F)
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
ng*day/mL | 7.82 (2.87) | 9.61 (3.20) | 11.08 (5.42) | 11.52 (7.92) | 18.20 (8.80) | 21.59 (15.15)

2. Primary Outcome: Maximum Change From Baseline for Neopterin for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of standard pharmacodynamic (PD) metric (maximal difference at a single time-point) for neopterin at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
ng/mL | 3.50 (1.06) | 4.22 (1.67) | 4.93 (1.85) | 3.17 (2.23) | 5.01 (2.10) | 5.87 (1.7)

3. Secondary Outcome: Area Under the Curve (AUC) for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of pharmacokinetic characteristic (AUC of free drug concentration) at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL*day
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
pg/mL*day | 99.4 (45) | 223 (46) | 386 (28) | 970 (44) | 2226 (37) | 2740 (65)

4. Secondary Outcome: Maximum Concentration (Cmax) for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of pharmacokinetic characteristic (Cmax) at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
pg/mL | 39.5 (54) | 90.8 (66) | 143 (33) | 191 (49) | 434 (49) | 509 (65)

5. Secondary Outcome: Area Under Effect Curve (AUEC) for Myxovirus-resistance Protein A (MxA) for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of standard PD metric (AUEC [baseline subtracted]) for MxA at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
ng*day/mL | 140 (63) | 172 (92) | 211 (102) | 458 (303) | 732 (591) | 1137 (592)

6. Secondary Outcome: Maximum Change From Baseline for Myxovirus-resistance Protein A (MxA) for Interferon Beta-1a and Peginterferon Beta-1a
Description: The values and variability of standard PD metric (maximal difference at a single time-point) for MxA at low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a
Time Frame: as for outcome 1
Population: Analysis population includes all subjects who did not discontinue before the end of study.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 12 | 11
ng/mL | 52.9 (28.7) | 62.9 (31.7) | 73.4 (35.5) | 86.7 (49.0) | 117.6 (73.0) | 175.5 (93.5)

7. Secondary Outcome: Pharmacodynamic Model Parameter, Emax (Maximum Effect), for Neopterin Area Under the Effect Curve Models With Interferon Beta-1a or Peginterferon Beta-1a
Description: Model parameter (Emax) for neopterin area under the effect curve models calculated after combining data from low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a with placebo data. As such, the placebo arm was included in both analyses.
Time Frame: as for outcome 1
Population: Analysis population for each group was limited to those subjects administered interferon beta-1a or placebo (interferon beta-1a group) or peginterferon beta-1a or placebo (peginterferon beta-1a group) who completed the study. One outlying result from peginterferon beta-1a high dose was excluded. Results from subjects administered placebo were used in all analyses. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 10000 repetitions.
Measure: Mean (95% Confidence Interval); unit: ng/mL*day
Groups:
- Interferon Beta-1a: Area Under the Effect Curve Model for Neopterin: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all interferon beta-1a and placebo arms.
- Peginterferon Beta-1a: Area Under the Effect Curve Model for Neopterin: Model-based analysis using individual subject baseline-subtracted area under the effect curve results from all peginterferon beta-1a and placebo arms.
Arm/Group | Interferon Beta-1a: Area Under the Effect Curve Model for Neopterin | Peginterferon Beta-1a: Area Under the Effect Curve Model for Neopterin
Number analyzed (Participants) | 47 | 46
ng/mL*day | 13.3 [9.3 to 19.3] | 44.0 [28.8 to 59.7]

8. Secondary Outcome: Pharmacodynamic Model Parameter, ED50 (Half Maximal Effect Dose), for Neopterin Area Under the Effect Curve Models With Interferon Beta-1a or Peginterferon Beta-1a
Description: Model parameter (ED50) for neopterin area under the effect curve models calculated after combining data from low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a with placebo data. As such, the placebo arm was included in both analyses.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: ug
Arm/Group | Interferon Beta-1a: Area Under the Effect Curve Model for Neopterin | Peginterferon Beta-1a: Area Under the Effect Curve Model for Neopterin
Number analyzed (Participants) | 47 | 46
ug | 4.5 [0.3 to 15.1] | 84.1 [30.8 to 422.0]

9. Secondary Outcome: Pharmacodynamic Model Parameter, Emax, for Neopterin Maximum Change From Baseline Models With Interferon Beta-1a or Peginterferon Beta-1a
Description: Model parameter (Emax) for neopterin maximum change from baseline models calculated after combining data from low, intermediate, and high doses of interferon beta-1a and peginterferon beta-1a with placebo data. As such, the placebo arm was included in both analyses.
Time Frame: as for outcome 1
Population: Analysis population for each group was limited to those subjects administered interferon beta-1a or placebo (the interferon beta-1a group) or administered peginterferon beta-1a or placebo (peginterferon beta-1a) who completed the study. Results from subjects administered placebo were used in all analyses. Confidence intervals for model parameters were generated using bootstrapping of the estimated model with 10000 repetitions.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Interferon Beta-1a: Maximum Change From Baseline Model for Neopterin: Model-based analysis using individual subject maximum change from baseline results from all interferon beta-1a and placebo arms.
- Peginterferon Beta-1a: Maximum Change From Baseline Model for Neopterin: Model-based analysis using individual subject maximum change from baseline results from all peginterferon beta-1a and placebo arms.
Arm/Group | Interferon Beta-1a: Maximum Change From Baseline Model for Neopterin | Peginterferon Beta-1a: Maximum Change From Baseline Model for Neopterin
Number analyzed (Participants) | 47 | 47
ng/mL | 5.7 [4.1 to 6.3] | 8.2 [5.7 to 12.4]

10. Secondary Outcome: Pharmacodynamic Model Parameter, ED50, for Neopterin Maximum Change From Baseline Models With Interferon Beta-1a or Peginterferon Beta-1a
Description: Model parameter (ED50) for neopterin maximum change from baseline models calculated after combining data from low, intermediate, and high doses of interferon beta-1a or peginterferon beta-1a with placebo data. As such, the placebo arm was included in both analyses.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: ug
Arm/Group | Interferon Beta-1a: Maximum Change From Baseline Model for Neopterin | Peginterferon Beta-1a: Maximum Change From Baseline Model for Neopterin
Number analyzed (Participants) | 47 | 47
ug | 4.8 [0.7 to 13.5] | 44.3 [14.5 to 135.4]

ADVERSE EVENTS:
Time Frame: 6 days for subjects in interferon beta-1a arms and 13 days for subjects in peginterferon beta-1a or placebo treatment arms
Arm/Group | Arm A: Interferon Beta-1a Low Dose | Arm B: Interferon Beta-1a Intermediate Dose | Arm C: Interferon Beta-1a High Dose | Arm D: Peginterferon Beta-1a Low Dose | Arm E: Peginterferon Beta-1a Intermediate Dose | Arm F: Peginterferon Beta-1a High Dose | Arm G: Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 7/12 | 10/12 | 7/12 | 9/12 | 11/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Interferon Beta-1a Low Dose (N=12) | Arm B: Interferon Beta-1a Intermediate Dose (N=12) | Arm C: Interferon Beta-1a High Dose (N=12) | Arm D: Peginterferon Beta-1a Low Dose (N=12) | Arm E: Peginterferon Beta-1a Intermediate Dose (N=12) | Arm F: Peginterferon Beta-1a High Dose (N=12) | Arm G: Placebo (N=12)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 8 (10) | 2 (2) | 5 (7) | 9 (14) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 4 (4) | 2 (3) | 5 (7) | 5 (7) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (4) | 5 (5) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sweating fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04183491/Prot_001.pdf
  • Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT04183491/SAP_002.pdf
  • Informed Consent Form (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT04183491/ICF_000.pdf